CLINICAL TRIAL: NCT00031746
Title: Effects of Dietary Soy on Biomarkers of Prostate Cancer: A Prospective Phase II Study
Brief Title: Soy Protein Supplement in Preventing Prostate Cancer in Patients With Elevated Prostate-Specific Antigen Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CALGB-79806; U10CA076001 (NIH); CALGB-79806; NCI-P02-0207; CDR0000069221 (Registry Identifier: NCI Physicians Data Query)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Soybean Proteins; alpha-casein-binding proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- soy protein + isoflavones (Active Comparator)
  Interventions: Dietary Supplement: soy protein isolate
- casein proteins (Active Comparator)
  Interventions: Dietary Supplement: casein proteins

INTERVENTIONS:
Dietary Supplement: soy protein isolate — 25 mg daily
  Arms: soy protein + isoflavones
Dietary Supplement: casein proteins — 25 mg daily
  Arms: casein proteins

SUMMARY:
RATIONALE: Soy protein supplement may prevent or delay the development of prostate cancer in patients who have elevated prostate-specific antigen (PSA) levels.

PURPOSE: Randomized phase II trial to determine the effectiveness of soy protein supplement in preventing prostate cancer in patients who have elevated PSA levels.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the reduction in the rate of prostatic cellular proliferation in patients with an elevated PSA (5 to 10 ng/mL) and a negative biopsy for prostate cancer when treated with daily soy protein supplements vs placebo.
* Compare the effect of these regimens on additional biomarkers of prostate cancer (PSA, high-grade prostate intraepithelial neoplasia, induction of apoptosis, sex steroid receptor expression, and loss of glutathione S-transferase-pi) in these patients.
* Compare the effect of these regimens on quality of life, including urinary and sexual function, in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to race (Caucasian vs African American). After 2 weeks of daily oral placebo, patients are randomized to 1 of 2 arms.

* Arm I: Patients receive oral soy protein supplement daily for 12 months.
* Arm II: Patients receive oral placebo daily for 12 months. Quality of life is assessed at baseline and at 6 and 12 months.

PROJECTED ACCRUAL: A total of 160 patients (80 per arm) will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed absence of prostate cancer

  * Atypical adenomatous hyperplasia or prostatic intraepithelial neoplasia (high-grade or low-grade) allowed
  * Abnormal baseline transrectal ultrasound and digital rectal exam allowed
  * Biopsy may be before or after study entry, but must be within the past 90 days
* PSA 5-10 ng/mL

PATIENT CHARACTERISTICS:

Age:

* 50 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No known allergy to soy protein or milk protein
* No invasive cancer within the past 5 years except non-melanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No prior hormonal therapy
* No prior finasteride
* No concurrent hormonal therapy
* No concurrent finasteride

Radiotherapy:

* Not specified

Surgery:

* At least 6 months since prior transurethral resection of the prostate
* No prior orchiectomy
* No concurrent orchiectomy

Other:

* No other concurrent soy products

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2000-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Reduction of prostatic cellular proliferation rates by 50% as measured by Ki-67 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James L. Mohler, MD, Study Chair — Roswell Park Cancer Institute
Locations (5):
- United States (5):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - Community General Hospital of Greater Syracuse, Syracuse, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio